CLINICAL TRIAL: NCT07335172
Title: Bedside Gastric Ultrasound Before Elective Cesarean Section: Observational Study
Brief Title: Gastric Ultrasound Before Elective Cesarean Section
Status: Not yet recruiting | Type: Observational
Sponsor: Ekin Deniz KUTLU (Other)
Responsible Party: Sponsor-Investigator, Ekin Deniz KUTLU, Anesthesiology and Reanimation researcher/ Doctor, Gazi University
Organization: Gazi University (Other)
Other Study IDs: 218
Record Dates: First submitted 2026-01-05; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-11

CONDITIONS: Gastric Ultrasound; Elective Cesarean Section; Pregnant Women
Keywords: Gastric Ultrasound; elective cesarean section

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ASA II term pregnant women aged 18-45 years scheduled for elective cesarean delivery

SUMMARY:
Due to the physiologically delayed gastric emptying in pregnant women, the potential risk of aspiration before cesarean delivery constitutes an important source of perioperative complications, and when it occurs, it is associated with increased maternal morbidity and/or mortality. Systematic reviews and meta-analyses have demonstrated that, compared with non-pregnant women, gastric emptying is delayed particularly during the first trimester of pregnancy, and that gastric emptying does not occur in cases who have consumed solid food within the last 8 hours and in whom labor has begun.

This study aims to evaluate preoperative gastric volumes by ultrasonography in ASA II pregnant women (according to the American Society of Anesthesiologists classification, healthy parturients without complications) scheduled to undergo elective cesarean delivery under general or spinal anesthesia, based on different fasting durations for solid and liquid intake, with the type of liquid.

Although previous research in pregnant populations has predominantly focused on the importance of gastric ultrasonography in the presence of gestational diabetes mellitus, this thesis study aims to generate data from the general population. The findings are expected to enable individualized preventive measures to reduce aspiration-related complications during cesarean deliveries performed under general or spinal anesthesia, thereby contributing to patient safety.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-45 years
* Term pregnant women classified as ASA II scheduled for elective cesarean section
* Those who voluntarily agree to participate in the study

Exclusion Criteria:

* Cases requiring emergency (Lucas classification based on the urgency of caesarean section, Category 1-2)
* Multiple pregnancies

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: Healthy term pregnant women aged 18-45 years, ASA II, scheduled for elective cesarean section
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Obstetric Ultrasonographic Assessment: Gastric volume | 60-90 minutes before surgery
  1. Obstetric Ultrasonographic Assessment: Gastric Volume
  Gastric volume will be calculated by ultrasonography (with two mathematical models from the literature) before elective cesarean delivery and recorded in milliliters.
Time of last solid food / liquid intake The time of the last solid food and liquid intake by the pregnant women will be recorded in hours. Liquid type will be also recorded. | 60-90 minutes before surgery
  The time of the last solid food and liquid intake by the pregnant women will be recorded in hours. Liquid type will be also recorded.

SECONDARY OUTCOMES:
Preoperative data | 60-90 minutes before surgery
  In the preoperative period; the patient's age, weight (kg), body mass index (BMI, kg/m²), and gestational age (weeks + days) will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Ekin KUTLU, Principal Investigator — Gazi University Hospital

IPD SHARING:
Plan to Share IPD: No